CLINICAL TRIAL: NCT04888949
Title: An Phase2 Study of ADR-001 in Patients With Severe Pneumonia Caused by SARS-CoV-2 Infection
Brief Title: A Study of ADR-001 in Patients With Severe Pneumonia Caused by SARS-CoV-2 Infection (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rohto Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADR-001-1921
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2 Infection( COVID-19 )

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell (Experimental): 4 times dose of Mesenchymal stem cell
  Interventions: Biological: Mesenchymal stem cell
- Placebo (Placebo Comparator): Saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Mesenchymal stem cell — 1*10^8 cells are administered once a week, total four times intravenously.
  Arms: Mesenchymal stem cell
Biological: Placebo — Commercially available saline.
  Arms: Placebo

SUMMARY:
Safety and efficacy of ADR-001 are evaluated in Patients with Severe Pneumonia caused by SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Patients with Severe Pneumonia caused by SARS-CoV-2 infection are enrolled to the study. Adipose-derived mesenchymal stem cells (AD-MSCs) are administered once a week, total four times intravenously. Safety and efficacy of AD-MSCs are evaluated for 12 weeks after first administer.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection is confirmed on antigen test or PCR test
* Pulmonary infiltrative shadow is confirmed on chest X-ray test
* PaO2/FiO2 <=200mmHg at the time of screening

Exclusion Criteria:

* Continue treatment for Pneumonia before SARS-CoV-2 infection
* SOFA score >= 15
* Infection type on DIC diagnosis criteria >= 4
* Deep Venous Thrombosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Ventilator Free Days | Day 28
  Ventilator Free Days which appear in subjects with ADR-001 treatment are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Okawa Sumito, Study Director — Rohto Pharmaceutical Co., Ltd.
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan